CLINICAL TRIAL: NCT03631654
Title: Ivabradine in Stage D Heart Failure Patients on Chronic Inotropes: A Pilot Study
Brief Title: Ivabradine in Stage D Heart Failure Patients on Chronic Inotropes
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to obtain funding
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Stephen Gottlieb, Professor of Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HP-00080414
Record Dates: First submitted 2018-08-03; First posted 2018-08-15 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure NYHA Class IV
MeSH Terms: interventions — Ivabradine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Drug: Placebos
- Intervention (Experimental)
  Interventions: Drug: Ivabradine

INTERVENTIONS:
Drug: Ivabradine — Ivabradine administration--tablets given 5 mg twice daily for 2 weeks, then 7.5 mg twice daily
  Arms: Intervention
Drug: Placebos — Placebo
  Arms: Control

SUMMARY:
Ivabradine, a selective inhibitor of the If current in the sinoatrial node, provides heart rate reduction and leads to a reduction in heart failure hospitalizations. For this reason, the American College of Cardiology (ACC) and the American Heart Association (AHA) guidelines provide a class IIa recommendation for ivabradine in stable heart failure patients with LVEF 35% and New York Heart Association (NYHA) class II-III symptoms who are on a beta blocker at maximum tolerated dose with a resting heart rate of 70 beats per minute or greater. While ivabradine leads to improvement in outcomes in stable NYHA class II-III chronic heart failure patients, its role in class IV, stage D heart failure, and cardiogenic shock is less clear.

Ivabradine's effect on acute cardiogenic shock has been evaluated by two recent studies. In the MODIFY trial, a randomized control study evaluating ivabradine in patients with multiorgan dysfunction, the addition of ivabradine did not result in significant heart rate reductions or other positive clinical outcomes. However, a small prospective trial demonstrated a significant decrease in heart rate and NT-proBNP with the addition of ivabradine in patients with acute cardiogenic shock on dobutamine. While few data investigate ivabradine's role in acute cardiogenic shock, it has yet to be studied in heart failure patients on long-term inotropic therapy. Inotropes such as dobutamine and milrinone result in tachycardia and may lead to ventricular arrhythmias. Moreover, patients on chronic inotropes are typically off beta blockers and have few pharmacological options available to help reduce heart rates. Ivabradine may have a role in decreasing heart rate and improving outcomes in patients on chronic inotropes.

Given the benefits of ivabradine in stable chronic heart failure patients, we plan to perform a study investigating the role of ivabradine in NYHA Stage D patients on home inotropes.

Our primary objective is to analyze changes in two cardiac biomarkers, NT-proBNP and high-sensitivity troponin. Our secondary outcomes include changes in noninvasive echocardiographic hemodynamics, changes in arrhythmia burden, and heart failure symptom modification based on 6-minute walk test results.

ELIGIBILITY:
Inclusion Criteria:

* NYHA Stage D heart failure on 2 weeks of consecutive IV dobutamine or milrinone
* Followed at UMMC outpatient heart failure clinic or admitted to advanced heart failure inpatient service and planning to follow up at UMMC outpatient heart failure clinic

Exclusion Criteria:

* Patients who are already on ivabradine
* Patients who are not willing to follow-up with UMMC outpatient heart failure team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Cardiac biomarkers | One month
  NT-pro BNP and high sensitivity troponin

SECONDARY OUTCOMES:
Echocardiogram | 2 weeks, and one month
  ejection fraction (%)
6-minute walk test | 2 weeks, and one month
  Distance walked (meters) in 6 minutes